CLINICAL TRIAL: NCT06979544
Title: A Randomized, Blinded, Placebo-Controlled Study to Evaluate the Saftey and Efficacy of Oral LPCN 1154A in Women With Postpartum Depression
Brief Title: A Study to Assess the Safety and Efficacy of Oral LPCN 1154A in Women With Severe PPD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPCN 1154-24-002a
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Depression, Postpartum; Depression, Post-Partum; Postpartum Depression (PPD); Post-Natal Depression; Peripartum Depression; Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LPCN 1154A Tablets (Experimental): LPCN 1154A
  Interventions: Drug: LPCN 1154A
- Placebo Tablets (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LPCN 1154A — Oral LPCN 1154A tablets for 48 hours
  Other Names: Brexanolone
  Arms: LPCN 1154A Tablets
Drug: Placebo — Oral Placebo Tablets for 48 hours
  Arms: Placebo Tablets

SUMMARY:
The purpose of this research study is to test the study drug, LPCN 1154A, as a possible treatment for postpartum depression (PPD). The trial aims to determine:

* If LPCN 1154A reduces depressive symptoms in subjects with severe PPD
* How well LPCN 1154A is tolerated and what side effects it may cause
* If LPCN 1154A reduces anxiety symptoms in subjects with severe PPD

ELIGIBILITY:
Key Inclusion Criteria:

* Are female between 15 and 45 years of age, inclusive;
* Have had a depressive episode that began no earlier than third trimester and later than the first 4 week following delivery
* Are < 12 months postpartum at Screening
* Hamilton Depression Rating Scale (HAM-D) 17-item score indicative of severe depression

Key Exclusion Criteria:

* Have a history of bipolar disorder, schizophrenia or schizoaffective disorder
* Are currently experiencing active psychosis per Investigator assessment
* Have a history of suicidal behavior within 1 year
* Have a history of seizure within 6 months of Screening

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HAM-D17 total score compared to placebo | Baseline to Hour 60
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) contains 17 individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia (initial, middle, and late), work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic and somatic), gastrointestinal symptoms, general somatic symptoms, sexual interest, hypochondriasis, insight, and weight loss. The total score ranges from 0 to 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Incidence, severity, and causality of AEs and SAEs | upto Day 30
  Adverse events (AEs) and Serious Adverse Events (SAEs)
Change from baseline in HAM-D17 total score | Baseline at Hours 12, and 36, Day 7 and Day 30
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) evaluates mood, suicide, work and interests, retardation, agitation, gastrointestinal symptoms, somatic symptoms, hypochondriasis, body weight and insight The total score ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17 response | Baseline to Hours 12, and 36, 60, Day 7 and Day 30
  Defined as having a 50% or greater reduction from baseline in HAM-D17 total score. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17 remission | Hours 12, and 36, 60, Day 7 and Day 30
  Defined as having a HAM-D17 total score ≤7. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
Patient Global Impression - Change (PGI-C) scale positive response | Hours 12, and 36, 60, Day 7 and Day 30
  The PGI-C scale is a 7-point scale that ranges from "1-very much better" to "7-very much worse" that allows participants to self- report their perception of improvement or decline of overall symptoms since starting treatment.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) total score | Baseline to Hour 60 and Day 30
  The MADRS is a 10-item assessment that evaluates mood/thoughts, sleep, appetite, tension, concentration The total score ranges from 0 to 60, with higher scores indicating more severe depression.
Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) total score | Baseline to Hours 12, 36, 60 Day 7 and Day 30
  The HAM-A is a 14-item assessment that evaluates mood, tension, fear, memory/concentration, sleep, and physical symptoms affecting somatic, sensory, respiratory, cardiovascular, gastrointestinal, genitourinary, and autoimmune systems as it relates to anxiety. The total score ranges from 0 to 56, with higher scores indicating more severe anxiety.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Advanced Research Center, Anahiem, California
  - Alliance Research Institute, Canoga Park, California
  - MedOne Clinical Research, LLC, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - Atlanta Behavioral Research, Atlanta, Georgia
  - CenExel Research Center, Decatur, Georgia
  - CenExel Research Center, Savannah, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Cypress Medical Research Center, LLC, Kansas City, Kansas
  - Best Clinical Trials, New Orleans, Louisiana
  - Oasis Clinical Research, Las Vegas, Nevada
  - Monroe Biomedical Research, Monroe, North Carolina
  - Suburban Research Associates, Media, Pennsylvania
  - Gadolin Research, Beaumont, Texas
  - New Dawn Wellness and Medical Center, Houston, Texas
  - Maximos OB/GYN, League City, Texas
  - Populace Research, Provo, Utah

IPD SHARING:
Plan to Share IPD: No